CLINICAL TRIAL: NCT05951738
Title: Exposures to PRenatal and Postnatal Adverse Stressful Experiences: Multimodal Omics Signatures Underlying Stress Vulnerability and Resilience and as Novel Targets for Preventive Strategies.
Brief Title: Exposures to Perinatal Adverse Experiences: Multimodal Omics Signature of Stress Vulnerability and Resilience and Preventive Strategies
Acronym: PRESeNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Annamaria Cattaneo, Head of the Biological Psichiatry unit, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PRESeNT; 1749118 (Other Grant/Funding Number: FRRB - Fondazione Regionale per la Ricerca Biomedica)
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Perinatal Depression
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Depressed (Other)
  Interventions: Procedure: Blood and saliva collection; Behavioral: Psychometric scales; Other: Smartphone app
- At high risk (Other)
  Interventions: Procedure: Blood and saliva collection; Behavioral: Psychometric scales; Other: Smartphone app
- Control (Other)
  Interventions: Procedure: Blood and saliva collection; Behavioral: Psychometric scales; Other: Smartphone app

INTERVENTIONS:
Procedure: Blood and saliva collection — Blood and saliva samples from pregnant women; saliva samples from babies.
Behavioral: Psychometric scales — A battery of psychometric scales and questionnaires.
Other: Smartphone app — A smartphone application has been developed in the context of the study as a potential preventive and screening strategy.

SUMMARY:
The study aims at identifying:

1. specific biological and molecular alterations associated with development of depression in pregnancy or risk of it.
2. specific biological and molecular alterations due to exposure to maternal depression in utero that are still present in the offspring, that could possibly mediate the development of negative outcomes, and which are the possible clinical moderators of the associated risk;
3. whether antidepressant therapies prescribed by personal physician and the use of digital tools can have a preventive effect in the transmission of the risk from mothers to babies and in the development of depressive symptoms in high-risk pregnant women;

In order to achieve these, 80 pregnant women with depression, 80 at high-risk and 80 controls will be recruited and clinically monitored over pregnancy and postpartum along with their babies, specifically at these timepoints: 25th and 32nd weeks of gestation, 1 week postpartum, 4 weeks postpartum, 8 weeks postpartum, 12 months postpartum.

Women, based on their clinician choice, will receive antidepressants and will be provided with a smartphone app to monitor them, using a combination of personalised, daily self-reported assessments and sensors for passive data collection to cover mental and physical health.

Blood and saliva samples from pregnant women will be collected at the 25th and 32nd week of gestation to perform biological analyses.

Saliva samples from babies will be collected at 8 weeks and 12 months postpartum to perform biological analyses.

Clinical and psychological data will be collected from women at all timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of a singleton pregnancy
* Age ≥ 18 years

Exclusion Criteria:

* Uterine anomalies and obstetric complications
* Comorbidity with severe or chronic diseases
* Substance abuse
* Language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Differentially expressed genes and biological pathways modulation | 25th and 32nd weeks of gestation for pregnant women; 8 weeks and 12 months postpartum for babies.

SECONDARY OUTCOMES:
Rate and profile of DNA methylation | 25th and 32nd weeks of gestation for pregnant women; 8 weeks and 12 months postpartum for babies.
Cortisol levels | 25th and 32nd weeks of gestation for pregnant women; 8 weeks and 12 months postpartum for babies.
Immune-related factors levels | 25th and 32nd weeks of gestation for pregnant women; 8 weeks and 12 months postpartum for babies.
Smartphone app utility | From 25th of gestation to 12 months postpartum

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia
  - Centro Psiche Donna - Ospedale Macedonio Melloni - ASST Fatebenefratelli Sacco, Milan
  - Ospedale San Raffaele, Milan
  - ASST Bergamo ovest, Treviglio

IPD SHARING:
Plan to Share IPD: Undecided